CLINICAL TRIAL: NCT03292484
Title: A Multicenter, Open-Label, Longer-Term Study of AR101 Characterized Oral Desensitization Immunotherapy in Subjects Who Participated in a Prior AR101 Study
Brief Title: Longer-term Study of AR101 in Subjects Who Participated in a Prior AR101 Study (ARC008)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aimmune Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARC008
Record Dates: First submitted 2017-09-21; First posted 2017-09-25 (Actual); Results first posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-11

CONDITIONS: Peanut Allergy
Keywords: AR101; Characterized Peanut Allergen; OIT (oral immunotherapy); Peanut Allergy; Allergy; Peanut-Allergic Children; Peanut-Allergic Adults; Desensitization; CPNA (Characterized Peanut Allergen)
MeSH Terms: conditions — Peanut Hypersensitivity; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AR101 (Experimental): Eligible participants who participated in a prior AR101 study received or continued initial dose escalation, up-dosing, and maintenance of AR101 at 300 milligrams (mg) per day until discontinuation criteria was met (maximum exposure: 4.8 years).
  Interventions: Biological: AR101

INTERVENTIONS:
Biological: AR101 — AR101

SUMMARY:
The purpose of this study is to assess AR101's safety, tolerability and efficacy over an extended dosing period.

DETAILED DESCRIPTION:
This study is enrolling participants by invitation only. This is an open-label, international, longer-term extension study for eligible subjects who have participated in one of the Aimmune AR101 clinical studies.

ELIGIBILITY:
Key Inclusion Criteria:

* Prior participation in an Aimmune AR101 clinical study or any future clinical study that identifies ARC008 as a follow-on study option in the protocol
* Written informed consent and/or assent from subjects/guardians as appropriate
* Use of effective birth control by sexually active female subjects of childbearing potential

Key Exclusion Criteria:

* Did not complete a minimum of 3 months of AR101 maintenance therapy if the subject was assigned to AR101 in the parent study
* Currently receiving or received within 5 years prior to Screening any type of peanut or other food allergen immunotherapy, except AR101 or unless allowed in the parent study, and except during the follow-up observation period in this study
* Discontinued early from the parent study

Ages: 1 Year to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 911 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jen Garcia, Study Chair — Director, Clinical Operations
Locations (93):
- United States (65):
  - Alabama Allergy and Asthma Center, Birmingham, Alabama
  - Medical Research of Arizona, Allergy, Asthma & Immunology Associates, Scottsdale, Arizona
  - Banner Univ. of Arizona Medical Center, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Jonathan Corren, M.D., Inc., Los Angeles, California
  - Children's Hospital Los Angeles, Division of Clinical Immunology and Allergy, Los Angeles, California
  - Allergy & Asthma Associates of Southern California, Mission Viejo, California
  - Sean N. Parker Center for Allergy and Asthma Research LPCH El Camino Hospital, Mountain View, California
  - Stanford University, Palo Alto, California
  - Peninsula Research Associates, Rolling Hills Estates, California
  - Allergy & Asthma Medical Group and Research Center, San Diego, California
  - Rady Children's Hospital, Div. of Allergy & Immunology, San Diego, California
  - UCSF, Benioff Children's Hospital - Allergy and Immunology, San Francisco, California
  - Allergy & Asthma Associates of Santa Clara Valley Research Center, San Jose, California
  - UCLA Medical Center, Santa Monica, Santa Monica, California
  - Bay Area Allergy, Walnut Creek, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Asthma & Allergy Associates, Colorado Springs, Colorado
  - National Jewish Health, Denver, Colorado
  - Colorado Allergy & Asthma Centers, P.C., Denver, Colorado
  - Children's National Health System, Washington D.C., District of Columbia
  - Sher Allergy Specialists - Center for Cough, Largo, Florida
  - Allergy Associates of the Palm Beaches, North Palm Beach, Florida
  - Sarasota Clinical Research, Sarasota, Florida
  - University of South Florida, Asthma Allergy & Immunology Clinical Research Unit, Tampa, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Atlanta Allergy & Asthma Clinic, Marietta, Georgia
  - Idaho Allergy and Research, Eagle, Idaho
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - The University of Chicago Medicine, Comer Children's Hospital, Chicago, Illinois
  - Sneeze, Wheeze, & Itch Associates, Normal, Illinois
  - Riley Children's Specialists, Carmel, Indiana
  - Deaconess Clinic, Inc., Evansville, Indiana
  - Family Allergy & Asthma Research Institute, Louisville, Kentucky
  - Chesapeake Clinical Research, Inc., Baltimore, Maryland
  - Johns Hopkins Hospital, Pediatric Clinical Research Unit, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Univ. of Michigan Health System, Div. of Allergy and Clinical Immunology, Ann Arbor, Michigan
  - Clinical Research Institute Inc., Plymouth, Minnesota
  - Children's Mercy on Broadway, Kansas City, Missouri
  - Atlantic Research Center, Ocean City, New Jersey
  - Princeton Center for Clinical Research, Skillman, New Jersey
  - Northwell Health System, Great Neck, New York
  - Jaffe Food Allergy Institute Icahn School of Medicine at Mount Sinai, New York, New York
  - Univ. of Rochester Medical Center, Golisano Children's Hosp., Rochester, New York
  - University of North Carolina at Chapel Hill, Clinical & Translational Research Center, Chapel Hill, North Carolina
  - Clinical Research of Charlotte, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio
  - Oklahoma Institute of Allergy and Asthma Clinical Research, Oklahoma City, Oklahoma
  - Columbia Asthma & Allergy Clinic, Clackamas, Oregon
  - Baker Allergy, Asthma and Dermatology, Portland, Oregon
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - National Allergy and Asthma Research, LLC, North Charleston, South Carolina
  - Le Bonheur Children's Hospital, Outpatient Bldg., Memphis, Tennessee
  - 'Specially for Children Allergy, Asthma and Immunology Clinic, Austin, Texas
  - Specially for Children Allergy, Asthma and Immunology Clinic, Austin, Texas
  - Children's Health, Dallas, Texas
  - Western Sky Medical Research, El Paso, Texas
  - Texas Children's Hospital, Baylor College of Medicine, Houston, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - ASTHMA, Inc. Clinical Research Center, Seattle, Washington
- Canada (5):
  - McMaster University Medical Center, Hamilton, Ontario
  - Triple A Lab, Hamilton, Ontario
  - Cheema Research Inc., Mississauga, Ontario
  - Ottawa Allergy Research Corp, Ottawa, Ontario
  - Gordon Sussman Clinical Research, Toronto, Ontario
- France (4):
  - Unité de dermatologie Pédiatrique, Hôpital Pellegrin-Enfants, Bordeaux, Cedex
  - Hopital Saint Vincent de Paul- Service d'Allergologie, Lille, Cedex
  - Jeanne de Flandre Hospital -Paediatric Allergy and Pulmonology Center, Lille, Cedex
  - Service d'Allergologie Nouvel Hôpital Civil Hôpitaux Univesitaires de Strasbourg, Strasbourg, Cedex
- Germany (2):
  - Charité Universitaetsmedizin Berlin, Berlin
  - University of Frankfurt, Frankfurt
- Ireland (2):
  - Cork University Hospital, UCC Department of Paediatrics and Child Health, Cork
  - National Children's Research Centre, Our Lady's Children's Hospital Crumlin, Dublin
- Azienda Ospedaliera di Padova, Padua, Province Of Padua, Italy
- Netherlands (2):
  - Beatrix Children's Hospital, University Medical Center Groningen, Groningen
  - University Medical Center Groningen, Groningen
- Spain (3):
  - Hospital General Universitario Gregorio Marañón, Madrid
  - H. Infantil Universitario Niño Jesús, Servicio de Alergia, Madrid
  - Madrid Hospital Clinico San Carlos, Servicio de Alergia, Madrid
- Sachsska Children and Youth Hospital, Stockholm, Sweden
- United Kingdom (8):
  - Leicester Royal infirmary, Leicester, Leicestershire
  - James Paget University Hospital, Gorleston-on-Sea, Norfolk
  - Guy & St Thomas' NHS Foundation Trust, Children Allergies Department, London
  - St Mary's Hospital - Paediatric Research Unit, London
  - Children's Clinical Research Facility, Royal Manchester Children's Hospital, Manchester
  - Sheffield Children's Hospital, Sheffield
  - University Hospitals Southampton Foundation NHS Trust, Southampton
  - Central Manchester University Hospitals, Wythenshawe

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nilsson C, Scurlock AM, Dellon ES, Brostoff JM, Pham T, Ryan R, Brown KR, Adelman DC, Aceves SS. Onset of eosinophilic esophagitis during a clinical trial program of oral immunotherapy for peanut allergy. J Allergy Clin Immunol Pract. 2021 Dec;9(12):4496-4501. doi: 10.1016/j.jaip.2021.07.048. Epub 2021 Aug 11. No abstract available. PMID 34389504
- [Derived] Fernandez-Rivas M, Vereda A, Vickery BP, Sharma V, Nilsson C, Muraro A, Hourihane JO, DunnGalvin A, du Toit G, Blumchen K, Beyer K, Smith A, Ryan R, Adelman DC, Jones SM. Open-label follow-on study evaluating the efficacy, safety, and quality of life with extended daily oral immunotherapy in children with peanut allergy. Allergy. 2022 Mar;77(3):991-1003. doi: 10.1111/all.15027. Epub 2021 Sep 24. PMID 34320250

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 3, open-label study was conducted in participants who participated in a prior AR101 study at 89 investigational sites in 10 countries (Canada, France, Germany, Ireland, Italy, Netherlands, Spain, Sweden, United Kingdom, and the United States).
Pre-assignment Details: A total of 911 participants were enrolled in this study. After enrolling in ARC008, all participants received or continued initial dose escalation, up-dosing, and maintenance of AR101 at 300 milligrams (mg) per day.
Groups:
- AR101: Eligible participants who participated in a prior AR101 study received or continued initial dose escalation, up-dosing, and maintenance of AR101 at 300 mg per day until discontinuation criteria was met (maximum exposure: 4.8 years).
Period: Overall Study
Arm/Group | AR101
Started | 911
Safety Population (The safety population consisted of all participants who received AR101 during ARC008.) | 908
Participants Who Had an Open-label Food Challenge (OLFC) (At Month 12 and yearly thereafter, up to 58 months.) | 517
Participants Who Had a Double-blind, Placebo-Controlled Food Challenge (DBPCFC) (At end of treatment (Month 58).) | 211
Completed | 18
Not Completed | 893
Not completed — Participants did not have Disposition - Study Exit forms | 415
Not completed — Withdrew consent (unrelated to adverse event [AE]) | 86
Not completed — Protocol Violation | 2
Not completed — Investigator decision (unrelated to AE) | 13
Not completed — Sponsor decision | 349
Not completed — Lost to Follow-up | 7
Not completed — Coronavirus Disease 2019 | 1
Not completed — Other | 20

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all enrolled participants.
Arm/Group | AR101
Number analyzed (Participants) | 911
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.8 (4.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 359
  Male | 552
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38
  Not Hispanic or Latino | 842
  Unknown or Not Reported | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 106
  Black or African American | 18
  Native Hawaiian or Other Pacific Islander | 3
  White | 664
  Other | 65
  Multiple Races Reported | 53
  Not Collected | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An AE was any untoward medical occurrence in humans, whether or not considered related to the investigational product (IP), that occurred during the conduct of a clinical study. A SAE was any event that resulted in any of the following: death, life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions, congenital abnormality or birth defect, or important medical event that did not result in one of the above outcomes, but jeopardized the health of the study participant or required medical or surgical intervention to prevent one of the outcomes listed above. TEAEs were defined as those AEs with onset after the first dose of AR101 in ARC008 and no more than 30 days after the last dose of study drug.
Time Frame: From first dose of study drug through 30 days after last dose of study drug, up to 59 months
Population: The safety population consisted of all participants who received AR101 during ARC008.
Measure: Count of Participants; unit: Participants
Arm/Group | AR101
Number analyzed (Participants) | 908
Participants
  TEAEs | 866
  TESAEs | 42

2. Primary Outcome: Number of Participants With Premature Discontinuation of AR101 Dosing Due to TEAEs
Description: An AE was any untoward medical occurrence in humans, whether or not considered related to the IP, that occurred during the conduct of a clinical study. TEAEs were defined as those AEs with onset after the first dose of AR101 in ARC008 and no more than 30 days after the last dose of study drug.
Time Frame: From first dose of study drug through 30 days after last dose of study drug, up to 59 months
Population: The safety population consisted of all participants who received AR101 during ARC008.
Measure: Count of Participants; unit: Participants
Arm/Group | AR101
Number analyzed (Participants) | 908
Participants | 53

3. Primary Outcome: Number of Participants With Premature Discontinuation of AR101 Dosing Due to Chronic/Recurrent Gastrointestinal TEAEs
Description: An AE was any untoward medical occurrence in humans, whether or not considered related to the IP, that occurred during the conduct of a clinical study. TEAEs were defined as those AEs with onset after the first dose of AR101 in ARC008 and no more than 30 days after the last dose of study drug. Gastrointestinal (GI) AEs, typically chronic/recurrent GI AEs, that resulted in prolonged interruption of dosing are reported.
Time Frame: From first dose of study drug through 30 days after last dose of study drug, up to 59 months
Population: The safety population consisted of all participants who received AR101 during ARC008.
Measure: Count of Participants; unit: Participants
Arm/Group | AR101
Number analyzed (Participants) | 908
Participants | 25

4. Primary Outcome: Number of Participants With TEAEs That Led to a Change in Treatment Regimen
Description: An AE was any untoward medical occurrence in humans, whether or not considered related to the IP, that occurred during the conduct of a clinical study. TEAEs were defined as those AEs with onset after the first dose of AR101 in ARC008 and no more than 30 days after the last dose of study drug. Number of participants with TEAEs requiring dose interruption and dose reduction of study treatment are reported.
Time Frame: From first dose of study drug through 30 days after last dose of study drug, up to 59 months
Population: The safety population consisted of all participants who received AR101 during ARC008.
Measure: Count of Participants; unit: Participants
Arm/Group | AR101
Number analyzed (Participants) | 908
Participants
  TEAEs requiring dose interruption of study treatment | 669
  TEAEs requiring dose reduction of study treatment | 167

5. Primary Outcome: Number of Participants With TEAEs That Led to Early Withdrawal
Description: as for outcome 2
Time Frame: From first dose of study drug through 30 days after last dose of study drug, up to 59 months
Population: The safety population consisted of all participants who received AR101 during ARC008.
Measure: Count of Participants; unit: Participants
Arm/Group | AR101
Number analyzed (Participants) | 908
Participants | 27

6. Primary Outcome: Number of Participants Who Experienced a Treatment-emergent Anaphylactic Reaction
Description: Anaphylaxis was defined by a number of signs and symptoms that occurred alone or in combination within minutes up to a few hours after exposure to a provoking agent. Treatment-emergent anaphylactic reactions included anaphylactic reactions that occurred after first dose of AR101 in ARC008 through 30 days after last dose of study product but excluding anaphylactic reactions that occurred during or related to a food challenge.
Time Frame: From first dose of study drug through 30 days after last dose of study drug, up to 59 months
Population: The safety population consisted of all participants who received AR101 during ARC008.
Measure: Count of Participants; unit: Participants
Arm/Group | AR101
Number analyzed (Participants) | 908
Participants | 192

7. Primary Outcome: Number of Participants With Use of Epinephrine as a Rescue Medication
Description: Rescue medications were any medication used to treat individual acute allergic reactions during ARC008 and were according to recognized standards of care for allergy practice.
Time Frame: From first dose of study drug through 30 days after last dose of study drug, up to 59 months
Population: The safety population consisted of all participants who received AR101 during ARC008.
Measure: Count of Participants; unit: Participants
Arm/Group | AR101
Number analyzed (Participants) | 908
Participants | 234

8. Primary Outcome: Number of Participants Who Experienced Accidental or Non-accidental Food Allergy Episodes
Description: An accidental food allergen exposure was any known or suspected exposure to a food to which the participant was allergic, including peanut, whether or not it resulted in an AE. A non-accidental food allergen exposure was an intentional exposure to a food to which the participant was allergic, including peanut, whether or not it resulted in an AE. Treatment-emergent food allergy episodes included food allergy episodes that occurred after first dose of AR101 in ARC008 through 30 days after last dose of study product but excluding food allergy episodes that occurred during or related to a food challenge.
Time Frame: From first dose of study drug through 30 days after last dose of study drug, up to 59 months
Population: The safety population consisted of all participants who received AR101 during ARC008.
Measure: Count of Participants; unit: Participants
Arm/Group | AR101
Number analyzed (Participants) | 908
Participants
  Accidental Food Allergy Episodes | 208
  Non-accidental Food Allergy Episodes | 35

9. Primary Outcome: Number of Participants With TEAEs Following Accidental or Non-accidental Exposure to Peanut and Other Allergenic Foods
Description: An accidental food allergen exposure was any known or suspected exposure to a food to which the participant was allergic, including peanut, whether or not it resulted in an AE. A non-accidental food allergen exposure was an intentional exposure to a food to which the participant was allergic, including peanut, whether or not it resulted in an AE. An AE was any untoward medical occurrence in humans, whether or not considered related to the IP, that occurred during the conduct of a clinical study. Treatment-emergent food allergy episodes included food allergy episodes that occurred after first dose of AR101 in ARC008 through 30 days after last dose of study product but excluding food allergy episodes that occurred during or related to a food challenge.
Time Frame: From first dose of study drug through 30 days after last dose of study drug, up to 59 months
Population: The safety population consisted of all participants who received AR101 during ARC008.
Measure: Count of Participants; unit: Participants
Arm/Group | AR101
Number analyzed (Participants) | 908
Participants | 227

10. Primary Outcome: Number of Participants With Eosinophilic Esophagitis (EoE)
Description: EoE was diagnosed by biopsy/endoscopy.
Time Frame: From first dose of study drug through 30 days after last dose of study drug, up to 59 months
Population: The safety population consisted of all participants who received AR101 during ARC008.
Measure: Count of Participants; unit: Participants
Arm/Group | AR101
Number analyzed (Participants) | 908
Participants | 7

11. Secondary Outcome: Percentage of Participants Tolerating Each Challenge Dose in the Open-label Food Challenge (OLFC) and the Double-blind, Placebo-Controlled Food Challenge (DBPCFC)
Description: During the OLFC, single doses (300, 600, 1000, and 2000 mg) of peanut protein were conditionally tested using a food challenge mixture administered sequentially at 20- to 30-minute intervals. During the DBPCFC, single doses (3, 10, 30, 100, 300, 600, 1000, and 2000 mg) of peanut protein and placebo were conditionally tested using a food challenge mixture administered sequentially at 20- to 30-minute intervals up to a single highest challenge dose of 2000 mg.
Time Frame: OLFC: At Month 12 and yearly thereafter, up to 58 months; DBPCFC: End of treatment (Month 58)
Population: The safety population consisted of all participants who received AR101 during ARC008. Only those participants who had an OLFC or a DBPCFC are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | AR101
Number analyzed (Participants) | 517
percentage of participants
  OLFC: Tolerated a single highest dose of at least 300 mg | 98.6 [97.2 to 99.5]
  OLFC: Tolerated a single highest dose of at least 600 mg | 94.2 [91.8 to 96.1]
  OLFC: Tolerated a single highest dose of at least 1000 mg | 78.7 [74.9 to 82.2]
  OLFC: Tolerated a single highest dose of at least 2000 mg | 55.9 [51.5 to 60.2]
  DBPCFC: Tolerated a single highest dose of at least 3 mg: number analyzed (Participants) | 211
  DBPCFC: Tolerated a single highest dose of at least 3 mg | 100.0 [98.3 to 100.0]
  DBPCFC: Tolerated a single highest dose of at least 10 mg: number analyzed (Participants) | 211
  DBPCFC: Tolerated a single highest dose of at least 10 mg | 100.0 [98.3 to 100.0]
  DBPCFC: Tolerated a single highest dose of at least 30 mg: number analyzed (Participants) | 211
  DBPCFC: Tolerated a single highest dose of at least 30 mg | 99.5 [97.4 to 100.0]
  DBPCFC: Tolerated a single highest dose of at least 100 mg: number analyzed (Participants) | 211
  DBPCFC: Tolerated a single highest dose of at least 100 mg | 99.1 [96.6 to 99.9]
  DBPCFC: Tolerated a single highest dose of at least 300 mg: number analyzed (Participants) | 211
  DBPCFC: Tolerated a single highest dose of at least 300 mg | 94.8 [90.9 to 97.4]
  DBPCFC: Tolerated a single highest dose of at least 600 mg: number analyzed (Participants) | 211
  DBPCFC: Tolerated a single highest dose of at least 600 mg | 88.2 [83.0 to 92.2]
  DBPCFC: Tolerated a single highest dose of at least 1000 mg: number analyzed (Participants) | 211
  DBPCFC: Tolerated a single highest dose of at least 1000 mg | 75.8 [69.5 to 81.4]
  DBPCFC: Tolerated a single highest dose of at least 2000 mg: number analyzed (Participants) | 211
  DBPCFC: Tolerated a single highest dose of at least 2000 mg | 60.2 [53.2 to 66.8]

12. Secondary Outcome: Maximum Tolerated Challenge Dose at Each Food Challenge
Description: The maximum tolerated challenge dose for a food challenge was defined as the maximum single dose of peanut protein resulting in no more than mild symptoms and assessed by the investigator to have been tolerated (i.e., the participant did not experience any dose-limiting symptoms). During the OLFC, single doses (300, 600, 1000, and 2000 mg) of peanut protein were conditionally tested using a food challenge mixture administered sequentially at 20- to 30-minute intervals. During the DBPCFC, single doses (3, 10, 30, 100, 300, 600, 1000, and 2000 mg) of peanut protein and placebo were conditionally tested using a food challenge mixture administered sequentially at 20- to 30-minute intervals up to a single highest challenge dose of 2000 mg.
Time Frame: OLFC: At Month 12 and yearly thereafter, up to 58 months; DBPCFC: End of treatment (Month 58)
Population: as for outcome 11
Measure: Number; unit: mg
Arm/Group | AR101
Number analyzed (Participants) | 517
mg
  OLFC | 2000
  DBPCFC: number analyzed (Participants) | 211
  DBPCFC | 2000

13. Secondary Outcome: Number of Participants With Use of Epinephrine as a Rescue Medication During the Food Challenges
Description: Rescue medications were any medication used to treat individual acute allergic reactions during ARC008 and were according to recognized standards of care for allergy practice. During the OLFC, single doses (300, 600, 1000, and 2000 mg) of peanut protein were conditionally tested using a food challenge mixture administered sequentially at 20- to 30-minute intervals. During the DBPCFC, single doses (3, 10, 30, 100, 300, 600, 1000, and 2000 mg) of peanut protein and placebo were conditionally tested using a food challenge mixture administered sequentially at 20- to 30-minute intervals up to a single highest challenge dose of 2000 mg.
Time Frame: OLFC: At Month 12 and yearly thereafter, up to 58 months; DBPCFC: End of treatment (Month 58)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | AR101
Number analyzed (Participants) | 517
Participants
  OLFC | 110
  DBPCFC: number analyzed (Participants) | 211
  DBPCFC | 35

ADVERSE EVENTS:
Time Frame: From first dose of study drug through 30 days after last dose of study drug, up to 59 months
Description: The safety population consisted of all participants who received AR101 during ARC008.
Arm/Group | AR101
All-Cause Mortality (participants affected / at risk) | 0/908
Serious Adverse Events (participants affected / at risk) | 42/908
Other Adverse Events (participants affected / at risk) | 865/908
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AR101 (N=908)
Appendicitis (Infections and infestations) | 8 (8)
Croup infectious (Infections and infestations) | 2 (2)
Enterovirus infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
Meningitis viral (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1)
Salmonella bacteraemia (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 8 (8)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Coeliac disease (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Oral disorder (Gastrointestinal disorders) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 2 (2)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AR101 (N=908)
Nasopharyngitis (Infections and infestations) | 221 (474)
Upper respiratory tract infection (Infections and infestations) | 213 (421)
Viral infection (Infections and infestations) | 143 (250)
Influenza (Infections and infestations) | 108 (134)
COVID-19 (Infections and infestations) | 102 (114)
Gastroenteritis viral (Infections and infestations) | 90 (117)
Gastroenteritis (Infections and infestations) | 88 (118)
Rhinitis (Infections and infestations) | 76 (171)
Conjunctivitis (Infections and infestations) | 54 (79)
Pharyngitis streptococcal (Infections and infestations) | 54 (69)
Ear infection (Infections and infestations) | 50 (56)
Sinusitis (Infections and infestations) | 47 (60)
Vomiting (Gastrointestinal disorders) | 293 (769)
Abdominal pain (Gastrointestinal disorders) | 271 (2212)
Nausea (Gastrointestinal disorders) | 183 (1122)
Abdominal pain upper (Gastrointestinal disorders) | 173 (684)
Abdominal discomfort (Gastrointestinal disorders) | 166 (1028)
Diarrhoea (Gastrointestinal disorders) | 127 (272)
Oral pruritus (Gastrointestinal disorders) | 88 (739)
Lip swelling (Gastrointestinal disorders) | 68 (158)
Paraesthesia oral (Gastrointestinal disorders) | 59 (1215)
Lip pruritus (Gastrointestinal disorders) | 53 (253)
Dyspepsia (Gastrointestinal disorders) | 51 (173)
Cough (Respiratory, thoracic and mediastinal disorders) | 302 (949)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 169 (2368)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 165 (363)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 145 (317)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 118 (413)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 114 (272)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 107 (287)
Asthma (Respiratory, thoracic and mediastinal disorders) | 85 (160)
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 85 (466)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 60 (105)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 59 (131)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 50 (71)
Urticaria (Skin and subcutaneous tissue disorders) | 251 (862)
Pruritus (Skin and subcutaneous tissue disorders) | 191 (827)
Rash (Skin and subcutaneous tissue disorders) | 121 (182)
Eczema (Skin and subcutaneous tissue disorders) | 74 (143)
Erythema (Skin and subcutaneous tissue disorders) | 65 (125)
Pyrexia (General disorders) | 293 (597)
Illness (General disorders) | 61 (118)
Headache (Nervous system disorders) | 240 (816)
Anaphylactic reaction (Immune system disorders) | 187 (334)
Seasonal allergy (Immune system disorders) | 50 (87)
Eye pruritus (Eye disorders) | 83 (163)
Ear pain (Ear and labyrinth disorders) | 47 (65)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* Institutions cannot publish until the multi-center sponsor publication is published
* Or, institutions cannot publish until 18 months after study completion
* And Sponsor review of any publications is required prior to any institution publications according to contractual agreements

DOCUMENTS (2):
  • Study Protocol (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/84/NCT03292484/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-05): https://cdn.clinicaltrials.gov/large-docs/84/NCT03292484/SAP_001.pdf